CLINICAL TRIAL: NCT01544296
Title: Phase II Study of KHK6188 (A Placebo-controlled, Double Blind, Crossover Study of KHK6188 in Postherpetic Neuralgia)
Brief Title: A Comparative Study of KHK6188
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6188-004
Record Dates: First submitted 2012-02-21; First posted 2012-03-05 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- KHK6188, high dose (Experimental)
  Interventions: Drug: KHK6188
- KHK6188, low dose (Experimental)
  Interventions: Drug: KHK6188
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK6188
  Arms: KHK6188, high dose; KHK6188, low dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a placebo-controlled, double blind, crossover study to evaluate the efficacy and safety of KHK6188 in postherpetic neuralgia when administered orally for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain for ≥ 3 months and ≤ 1 year following onset of a herpes zoster rash
* Patients with a mean pain intensity score (11-point numerical rating scale) of ≥ 4
* Patients whose rash has been healed
* Patients who are able to fill their patient diary
* Patients who provided written voluntary informed consent to participate in the study

Exclusion Criteria:

* Patients who have other pain or disease which may impair the self assessment of pain
* Patients who have dementia, depression or schizophrenia which may affect the self assessment of pain
* History or presence of severe cardiovascular disease, hepatic dysfunction, renal failure, respiratory disease, blood disease or CNS disorder
* History or presence of a drug allergy
* Patients who have a history of a diagnosis of cancer or a treatment of cancer within 5 years prior to the study entry
* Patients received an investigational medication within 4 months (6 months for biologic medication such as antibody) prior to the informed consent
* Women of child bearing potential who do not agree to avoid pregnancy from the time of providing the consent until 3 months after the end of dosing, or men of reproductive potential who do not agree to avoid pregnancy from the time of the first dose until 3 months after the end of dosing
* Patients who are pregnant, lactating, or possibly pregnant
* Patients judged to be inappropriate to enter the study by a investigator or a subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change of pain intensity score | baseline and 2weeks

SECONDARY OUTCOMES:
Change of allodynia severity | baseline and 2 weeks
Change of global impression | baseline and 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Arakawa-ku, Tokyo, Japan